CLINICAL TRIAL: NCT04776941
Title: COVID-19: A Virtual Feasibility Study to Manage Stress
Brief Title: Expressive Writing for the Management of Stress in Cancer Survivors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020-0538; NCI-2021-00218 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0538 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-02-09; First posted 2021-03-02 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (questionnaires, messages, writing) (Experimental): Patients complete questionnaires over 30 minutes about their mood, health, and income at baseline, and 1, 3, and 6 months. Patients also read brief positive messages and write essays about their experiences over 30 minutes (non-stop) QW for 3 weeks.
  Interventions: Behavioral: Behavioral Intervention; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm II (questionnaires, messages, writing) (Active Comparator): Patients complete questionnaires over 30 minutes about their mood, health, and income at baseline, and 1, 3, and 6 months. Patients also read brief neutral messages and write essays about neutral topics over 30 minutes (non-stop) QW for 3 weeks.
  Interventions: Behavioral: Behavioral Intervention; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Behavioral: Behavioral Intervention — Read positive messages
  Other Names: Behavior Conditioning Therapy; Behavior Modification; Behavior or Life Style Modifications; Behavior Therapy; Behavioral Interventions; Behavioral Modification; Behavioral Therapy; Behavioral Treatment; Behavioral Treatments
  Arms: Arm I (questionnaires, messages, writing)
Behavioral: Behavioral Intervention — Write about positive experiences
  Other Names: Behavior Conditioning Therapy; Behavior Modification; Behavior or Life Style Modifications; Behavior Therapy; Behavioral Interventions; Behavioral Modification; Behavioral Therapy; Behavioral Treatment; Behavioral Treatments
  Arms: Arm I (questionnaires, messages, writing)
Behavioral: Behavioral Intervention — Write about neutral topics
  Other Names: Behavior Conditioning Therapy; Behavior Modification; Behavior or Life Style Modifications; Behavior Therapy; Behavioral Interventions; Behavioral Modification; Behavioral Therapy; Behavioral Treatment; Behavioral Treatments
  Arms: Arm II (questionnaires, messages, writing)
Behavioral: Behavioral Intervention — Read neutral messages
  Other Names: Behavior Conditioning Therapy; Behavior Modification; Behavior or Life Style Modifications; Behavior Therapy; Behavioral Interventions; Behavioral Modification; Behavioral Therapy; Behavioral Treatment; Behavioral Treatments
  Arms: Arm II (questionnaires, messages, writing)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Complete questionnaires

SUMMARY:
This clinical trial evaluates the effect of expressive writing for the management of stress in cancer survivors. Cancer diagnosis and treatment are associated with increased stress in cancer survivors related to concerns about family, career, relationships, finances, side effects of treatment, and death. This stress can be further exacerbated by social upheavals such as the COVID-19 pandemic. For safety reasons, many patients are isolated with restricted access to in-person health care and reduced social interaction with family and friends. Together with the economic uncertainties that come with this pandemic, these factors are likely to increase cancer survivors' stress levels. Expressive writing may provide a medium through which cancer survivors confront stressors and find meaning in their experience. The goal of this trial is to learn more about the experiences of cancer survivors during stressful times.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the feasibility of the virtual study for cancer survivors. II. To preliminarily assess the impact of the intervention for cancer survivors.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I (INTERVENTION): Patients complete questionnaires over 30 minutes about their mood, health, and income at baseline, and 1, 3, and 6 months. Patients also read brief positive messages and write essays about their experiences over 30 minutes (non-stop) once weekly (QW) for 3 weeks.

ARM II (CONTROL): Patients complete questionnaires over 30 minutes about their mood, health, and income at baseline, and 1, 3, and 6 months. Patients also read brief neutral messages and write essays about neutral topics over 30 minutes (non-stop) QW for 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Have a diagnosis of cancer within the past 3 years
* Are able to speak and read in English
* Have access to a computer or smart phone with internet connection
* All disease sites and all cancer stages are eligible for enrollment

Exclusion Criteria:

* Inability to provide informed consent
* Non-English speakers will be excluded because this is a feasibility study that will enroll only a limited number of participants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 414 (Estimated)
Dates: Start 2020-08-07 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Participant response rate | 1 month
Study completion rate | 1 month
Intervention adherence rate | 1 month

SECONDARY OUTCOMES:
Change in stress | Baseline and 1-, 3-, and 6-month follow-up
  Perceived stress will be measured with the 4-item Perceived Stress Scale. Scale scores range from 0-16, with low scores indicating low perceived stress and high scores indicating high perceived stress
Change in quality of life | Baseline and 1-, 3-, and 6-month follow-up
  Quality of life will be measured with the 7-item Functional Assessment of Cancer Therapy (FACT-G7). The items are rated on a 5-point scale from 0 - "not at all", to 4 - "very much". Scores range from 0-28, with higher scores indicating better quality of life.
Change in physical health (sleep, fatigue, and cancer related morbidities) | Baseline and 1-, 3-, and 6-month follow-up
  Sleep will be measured with the 19-item Pittsburgh Sleep Quality Index (PSQI). The PSQI global score ranges from 0 to 21, with a cut-off score of 5 or greater indicating poor sleep quality.
  Fatigue will be measured with the 4-item PROMIS Fatigue Short Form. This measure assesses the magnitude of fatigue in the past 7 days. Items are measured on a five-point scale (1= "not at all"; 5 = "very much") and summed. Higher scores indicate greater fatigue.
  Cancer related morbidities will be self-reported by participants and verified through medical record review.
  .
Change in psychological health (depressive symptoms, anxiety, and fear of cancer recurrence) | Baseline and 1-, 3-, and 6-month follow-up
  Depressive symptoms will be measured with the 4-item PROMIS Depression Short Form. This measure assesses the frequency of depressive symptoms in the past 7 days. Items are measured on a five-point scale (1= "never"; 5 = "always") and summed. Higher scores indicate more depressive symptoms.
  Anxiety will be measured with the 4-item PROMIS Anxiety Short Form. This measure assesses the frequency of anxiety in the past 7 days. Items are measured on a five-point scale (1= "never"; 5 = "always") and summed. Higher scores indicate greater anxiety.
  Fear of cancer recurrence will be measured with a single item added to the quality of life measure (F

CONTACTS AND LOCATIONS:
Overall Officials: Qian Lu, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org